CLINICAL TRIAL: NCT02416050
Title: Prospective Prediction of Cocaine Relapse After Inpatient Cessation by Combining Functional Imaging and Neuropsychological Biomarkers With Craving and Impulsivity Measures
Brief Title: Predicting Relapse After Cocaine Inpatient Cessation
Acronym: QUIT-COC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P120125; 2014-A01169-38 (Other: IDRCB)
Record Dates: First submitted 2015-02-02; First posted 2015-04-14 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Cocaine Dependence; Cocaine Use Disorder
Keywords: Cocaine; Dependence; Abstinence; Prediction; Model; Humans; MRI; Cognitive; Impulsivity; Craving
MeSH Terms: conditions — Cocaine-Related Disorders; Impulsive Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Brain MRI imagery — Brain MRI performed during the first week of inpatient cocaine cessation

SUMMARY:
Can brain MRI at entry of cocaine inpatient cessation attempt predict relapse during a three month follow-up ? Hypothesis : White matter losses in the prefrontal cortex are associated with relapse to cocaine use.

DETAILED DESCRIPTION:
A multivariate model using MRI parameters, craving score, impulsivity score, and neuropsychological testing results will be tested to predict relapse or continuous abstinence three month after cocaine inpatient cessation attempt.

ELIGIBILITY:
Inclusion Criteria:

* cocaine dependent patient requiring inpatient cessation
* 18 years old and older
* giving his/her consent to come back for visits up to three months
* having a social insurance

Exclusion Criteria:

* minor
* under guardianship
* restraint hospitalization
* contraindication to brain MRI
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cocaine dependent patient requiring inpatient cessation
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2015-02-03; Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
mean difference of fractional anisotropy of the prefrontal cortex (PFC) in patients abstinent from cocaine 3 months after inpatient detoxification compared to relapsers | at 3 months

SECONDARY OUTCOMES:
Comparisons between patients who remain abstinent from cocaine 3 months after inpatient detoxification and those who relapse | at baseline
  Differences in grey and white matter volumes : voxel-based morphometry (VBM) and in resting-state whole-brain activity default mode network (DMN)
Comparisons between patients who remain abstinent from cocaine 3 months after inpatient detoxification and those who relapse | at baseline
  Differences in scores of craving (visual scale and Obsessive compusilve craving scale (OCCS) questionnaire) and impulsivity (UPPS)
Comparisons between patients who remain abstinent from cocaine 3 months after inpatient detoxification and those who relapse | at baseline
  Differences in performance at the stroop test and in mental flexibility during an implicit set shifting task
Among abstinent patients who remain abstinent at three months only :Differences between baseline and 3 months measures of Diffusion Tensor Imagery (DTI), VBM and DMN | at 3 months
Among abstinent patients who remain abstinent at three months only: Differences in scores of craving (visual scale and OCCS questionnaire) and impulsivity (UPPS) | at 3 months
Among abstinent patients who remain abstinent at three months only: Differences in performance at the stroop test and in mental flexibility during an implicit set shifting task compared to baseline results | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence VORSPAN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Psychiatrie, Hôpital Fernand Widal, Paris, France